CLINICAL TRIAL: NCT06105502
Title: Systematic Evaluation of Psychotherapy Training: Impact of Supervision and Training on Student Learning and Patient Outcomes
Brief Title: Systematic Evaluation of Psychotherapy Training: Supervision, Student Learning, and Patient Outcomes
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-03668-01
Record Dates: First submitted 2023-08-25; First posted 2023-10-27 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Student Education
Keywords: psychotherapy; supervision; student learning; patient outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Psychotherapy students: The participating psychotherapy students will come from the following courses at the Center for Psychotherapy Education and Research: the psychotherapist program (six semesters), the specialist training for psychologists in adult psychiatry (six semesters), the basic training in evidence-based psychotherapeutic methods (three semesters), and the basic training in psychotherapy for residents in child, adolescent, and adult psychiatry (two semesters).
  Interventions: Behavioral: Psychotherapy education

INTERVENTIONS:
Behavioral: Psychotherapy education — Psychotherapy education, including supervision, lectures, and workshops

SUMMARY:
The project is a longitudinal observation study that aims to systematically evaluate selected parts of the material collected within the framework of the psychotherapy training conducted at the Center of Psychotherapy Education and Research unit at Karolinska Institutet and Region Stockholm, Sweden. Students at the unit, patients being administered psychotherapy by the students, and supervisors will participate in the study.

The aim of the present study is to investigate the associations between (1) content and quality of psychotherapy supervision, (2) student therapists' competence, and (3) patient outcomes following student-led psychotherapy.

DETAILED DESCRIPTION:
The project is a longitudinal observation study that aims to systematically evaluate selected parts of the material collected within the framework of the psychotherapy training conducted at the Center of Psychotherapy Education and Research unit at Karolinska Institutet and Region Stockholm, Sweden, from 2023 - 2028. The courses/programs that will be included in the project are the psychotherapist program (six semesters), the specialist training for psychologists in adult psychiatry (six semesters), the basic training in evidence-based psychotherapeutic methods (three semesters), and the basic training in psychotherapy for residents in child, adolescent, and adult psychiatry (two semesters). The element of the programs that will be evaluated is student-led psychotherapy, in which students conduct psychotherapy with patients in the public health care system.

The study's research subjects are supervisors, students, and their patients from the unit's student-led psychotherapies. Data consists of material that the supervisors and students have collected within the framework of the educational setting; the data are placed and stored on a secure digital platform (BASS). For objective estimates, the project also intends to code selected audio-recorded psychotherapy and supervision sessions.

The primary research questions are:

1. Do psychotherapy students' general and specific psychotherapy competence increase over time during training?
2. Can statistically significant and/or clinically meaningful patient improvements be observed after student-led psychotherapy?
3. Is students' psychotherapy competence significantly associated with patient outcomes?
4. Are aspects (content and quality) of the psychotherapy supervision setting significantly related to improved student therapists' competence?

The project also aims to psychometrically evaluate (validity and reliability) some of the included instruments.

ELIGIBILITY:
Inclusion Criteria:

* Students at one of the following courses/programs: Primary training in evidence-based psychotherapeutic methods (three semesters) and specialty trainee (ST) for doctors in child, adolescent, and adult psychiatry (two semesters), the postgraduate psychotherapist program (six semesters), and the specialist training program for clinical psychologists (six semesters).
* Clinical supervisors for the students in the abovementioned courses/programs.
* Patients in psychotherapy with students in the abovementioned courses/programs as therapists. The patients are regular patients at public health care facilities in psychiatry and primary care.
* Students, supervisors, and patients must consent to inclusion.

Exclusion Criteria:

* No exclusion criteria are applied.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Psychotherapy students at the Center for Psychotherapy Education and Research, Karolinska Institutet and Region Stockholm, Sweden
Sampling Method: Non-Probability Sample
Enrollment: 417 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
The Generalized Anxiety Disorder Assessment 7 (GAD-7) | Change from pre-treatment to immediately after the end of psychotherapy
  The GAD-7 is originally a measure for generalized anxiety disorder, but it is also frequently used to assess general anxiety. The form consists of seven items with a four-point scale. The range is 0-21 points. An eight item describes how disruptive the anxiety is from not at all to very significant, which is not included in the total score. The GAD-7 has been translated into Swedish and has shown good psychometric properties in terms of both reliability and validity.
The Patient Health Questionnaire-9 (PHQ-9) | Change from pre-treatment to immediately after the end of psychotherapy
  The PHQ-9 is a well-established depression questionnaire consisting of nine items that correspond to the diagnostic criteria for a major depressive episode according to the DMS-5. How often the symptoms have bothered the patient in the past two weeks is rated by the patient, at the start and end of treatment, on a four-point scale. The range is 0-27 points. The PHQ-9 has been translated into Swedish and has good internal consistency and test-retest reliability.
The WHO Disability Assessment Schedule (WHODAS 2.0) | Change from pre-treatment to immediately after the end of psychotherapy
  The WHODAS 2.0 is a widely used generic assessment instrument that provides a standardized method for measuring health and disability across cultures. The form is based on a set of questions from the International Classification of Functioning, Disability, and Health (ICF) that are sufficiently reliable and sensitive to measure changes after interventions. The form is available in seven different versions with 36 questions, 12 questions, and 12+24 questions as interview-administered, self-administered, and proxy-administered, respectively. In the project, the self-administered 12-question form is used.
The Alcohol Use Disorders Identification Test (AUDIT) | Change from pre-treatment to immediately after the end of psychotherapy for those patients scoring above the cut-off at pre-treatment
  The AUDIT is a widely used instrument for identifying hazardous and harmful alcohol consumption. The instrument was initially developed by the WHO and consists of a ten-item questionnaire designed to measure three domains: consumption, dependence, and alcohol-related harm. The project uses a cut-off point of 5 points as an indication of mild alcohol use disorder. The project uses the AUDIT-C, which includes the first three questions of the AUDIT.
The Sleep Condition Indicator (SCI) | Change from pre-treatment to immediately after the end of psychotherapy
  The SCI will be used to measure sleep disorders. The SCI contains eight questions regarding nocturnal symptoms, function, performance, duration, frequency, and severity. The form is translated into Swedish, and the psychometric properties have been shown in studies to be acceptable to good.
The Liebowitz Social Anxiety Scale, self-report (LSAS-SR) | Change from pre-treatment to immediately after the end of psychotherapy
  The LSAS-SR is only used for patients with social anxiety disorder or similar.
The Panic Disorder Severity Scale - Self-rated (PDSS-SR) | Change from pre-treatment to immediately after the end of psychotherapy
  The PDSS-SR is only used for patients with panic disorder or similar.
The Penn State Worry Questionnaire (PSWQ) | Change from pre-treatment to immediately after the end of psychotherapy
  The PSWQ is only used for patients with generalized anxiety disorder or similar.
The Posttraumatic Stress Disorder Checklist, version 5 (PCL-5) | Change from pre-treatment to immediately after the end of psychotherapy
  The PCL-5 is only used for patients with posttraumatic stress disorder or similar.
The Obsessive Compulsive Inventory-Revised (OCI-R) | Change from pre-treatment to immediately after the end of psychotherapy
  The OCI-R is only used for patients with obsessive-compulsive disorder or similar.
The Perceived Stress Scale-10 (PSS-10) | Change from pre-treatment to immediately after the end of psychotherapy
  The PSS-10 is only used for patients with stress or burnout problems or similar.
The Short Health Anxiety Inventory-14 (SHAI-14) | Change from pre-treatment to immediately after the end of psychotherapy
  The SHAI-14 is only used for patients with health anxiety problems or similar.
The Eating Disorder Examination Questionnaire (EDE-Q) | Change from pre-treatment to immediately after the end of psychotherapy
  The EDE-Q is only used for patients with eating disorders or similar.
The Drug Use Disorders Identification Test (DUDIT) | Change from pre-treatment to immediately after the end of psychotherapy
  The DUDIT is only used for patients with drug problems or similar.

OTHER OUTCOMES:
Psychotherapy summary | Student and patient data immediately after the end of psychotherapy
  At the end of each treatment, all students write a summary of the treatment consisting of questions about the student (socio-demographic and contextual), the patient (socio-demographic and clinical), and the treatment (e.g., content, duration, and compliance). The summary concludes by summarizing the results of the patient's pre- and post-measurements, which are guided by the patient's problem domain.
Cognitive Therapy Scale-Revised (CTS-R) | At first session, first treatment session, fifth treatment session, and last treatment session
  The CTS-R is a standard instrument for assessing CBT competence that measures both general psychotherapy aspects and specific CBT aspects. The instrument contains twelve items, which are rated on a scale from 0 to 6 points corresponding to six different categories of therapist competence (incompetent, novice, advanced, beginner, competent, knowledgeable, and expert). The CTS-R has been translated into Swedish and has shown acceptable psychometric properties in several studies.
Supervision Adherence and Guidance Evaluation (Short-SAGE) | At first session, first treatment session, fifth treatment session, and last treatment session
  The Short-SAGE is an observational tool to evaluate supervisors' skills and adherence to CBT supervision. Short-SAGE describes 14 behaviors (competencies of the supervisor and supervisee), grouped on two main factors: the Supervisor's set (specific behaviors of the supervisor that are believed to facilitate optimal learning through experience) and the Supervisee's set (specific learning competencies that can be observed in the supervisee). The assessor observes a tutoring session and rates the competencies observed on a 7-point scale. For training purposes, a simpler 3-point scale is used. The instrument is available in Swedish and English, is fairly new, and has only undergone preliminary psychometric evaluations.
Evaluation of Supervisory Skills and Adherence, 2019 (ESSA-19) | At first session, first treatment session, fifth treatment session, and last treatment session
  The ESSA-19 is a behavioral coding system to evaluate supervisors' skills and adherence to MI supervision. ESSA has been developed to be used as a tool for structured feedback to MI supervisors and as a measure of supervisory integrity in clinical trials. The manual has been developed at the unit 2019. The instrument is relatively new and has only undergone preliminary psychometric evaluations.
Supervision evaluation | At the middle of the student term (week 10 out of 20)
  A unit-developed set of 10 questions focusing on how the students perceive the supervisor and the supervision setting, e.g., regarding feedback, skills training, and activity.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Beckman, PhD, Principal Investigator — Center for Psychiatry Research, Karolinska Institutet and Region Stockholm
Locations (1):
- Center for Psychiatry Research, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
There is no ethical approval in place to allow for sharing IPD.